CLINICAL TRIAL: NCT02733536
Title: C-MAC Compared to Direct Laryngoscopy in Patients With Immobilized Cervical Spine by Unexperienced Physicians: A Randomized Crossover Manikin Trial
Brief Title: Intubation During Spinal Immobilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Principal Investigator, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23.01.2017.IRB
Record Dates: First submitted 2016-04-05; First posted 2016-04-11 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Endotracheal Intubation
Keywords: endotracheal intubation; trauma; paramedic
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Scenario A (Experimental): manikin with normal standard airway
  Interventions: Device: Standard endotracheal tube; Device: C-MAC
- Scenario B (Experimental): Cervical immobilization using a standard Patriot cervical extraction collar (Oessur Americas, Foothill Ranch, CA, USA), applied to the manikin's neck by an instructor.
  Interventions: Device: Standard endotracheal tube; Device: C-MAC
- Scenario C (Experimental): Cervical immobilization using a vacuum mattress (Ferno-Washington, Inc. Wilmington, OH, USA), applied to the manikin's neck by an instructor
  Interventions: Device: Standard endotracheal tube; Device: C-MAC

INTERVENTIONS:
Device: Standard endotracheal tube — 1) Direct laryngoscopy using a Macintosh laryngoscope with size 3 blade (Mercury Medical, Clearwater, FL, USA) with a conventional 7.0 mm internal diameter (ID) tracheal tube
Device: C-MAC — C-MAC introduced with a h size 3 blade.

SUMMARY:
The aim was to evaluate the performance of the C-MAC compared with Macintosh when performed in patients with immobilized cervical spine by unexperienced physicians.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* limited experience (<5 intubations) with "real-life" intubation using direct laryngoscopy
* novice phhysicians

Exclusion Criteria:

* not meet the above criteria
* practice with any videolaryngoscopy
* wrist or low back diseases
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Time required for successful intubation | 1 day

SECONDARY OUTCOMES:
success rate of intubation attempt | 1 day
  success rate of first intubation attempt
Cormack&Lehane grade | 1 day
  glottic view during intubation rate using Cormack&Lehane grade
Dental Compression | 1 day
  the severity of the potential dental trauma was calculated based on previously described modified grading scale (Svoldelli, 2009)
Ease of intubation | 1 day
  To access subjective opinion about the difficulty of each intubation method, participants were asked to rate it on a visual analog scale (VAS) with a score from 1 (extremely easy) to 10 (extremely difficult).

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Szarpak, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Department of Emergency Medicine, Warsaw, Masovia, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Truszewski Z, Szarpak L, Smereka J, Kurowski A, Evrin T, Czyzewski L. Comparison of the VivaSight single lumen endotracheal tube and the Macintosh laryngoscope for emergency intubation by experienced paramedics in a standardized airway manikin with restricted access: a randomized, crossover trial. Am J Emerg Med. 2016 May;34(5):929-30. doi: 10.1016/j.ajem.2016.02.054. Epub 2016 Feb 27. No abstract available. PMID 26979260
- [Background] Bogdanski L, Truszewski Z, Kurowski A, Czyzewski L, Zasko P, Adamczyk P, Szarpak L. Simulated endotracheal intubation of a patient with cervical spine immobilization during resuscitation: a randomized comparison of the Pentax AWS, the Airtraq, and the McCoy Laryngoscopes. Am J Emerg Med. 2015 Dec;33(12):1814-7. doi: 10.1016/j.ajem.2015.09.005. Epub 2015 Sep 21. PMID 26494629
- [Background] Gawlowski P, Smereka J, Madziala M, Szarpak L, Frass M, Robak O. Comparison of the Macintosh laryngoscope and blind intubation via the iGEL for Intubation With C-spine immobilization: A Randomized, crossover, manikin trial. Am J Emerg Med. 2017 Mar;35(3):484-487. doi: 10.1016/j.ajem.2016.11.064. Epub 2016 Nov 30. PMID 28041757
- [Derived] Karczewska K, Szarpak L, Smereka J, Dabrowski M, Ladny JR, Wieczorek W, Robak O, Frass M, Ahuja S, Ruetzler K. ET-View compared to direct laryngoscopy in patients with immobilized cervical spine by unexperienced physicians: A randomized crossover manikin trial. Anaesthesiol Intensive Ther. 2017;49(4):274-282. doi: 10.5603/AIT.a2017.0047. Epub 2017 Sep 27. PMID 28953308
- [Derived] Truszewski Z, Krajewski P, Fudalej M, Smereka J, Frass M, Robak O, Nguyen B, Ruetzler K, Szarpak L. A comparison of a traditional endotracheal tube versus ETView SL in endotracheal intubation during different emergency conditions: A randomized, crossover cadaver trial. Medicine (Baltimore). 2016 Nov;95(44):e5170. doi: 10.1097/MD.0000000000005170. PMID 27858851